CLINICAL TRIAL: NCT03992729
Title: Post-authorization Safety Study for Assessment of Pregnancy Outcomes in Patients Treated With Tildrakizumab
Brief Title: Safety Study for Prospective Assessment of Pregnancy Outcomes in Patients Treated With Tildrakizumab
Status: Recruiting | Type: Observational
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: TILD 3357-2
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tildrakizumab-Exposed Cohort: Exposure to tildrakizumab for the treatment of an approved indication
  Interventions: Drug: Pregnant women exposed to tildrakizumab
- Disease-Matched Comparison Cohort: No exposure to tildrakizumab at any time in the current pregnancy
  Interventions: Drug: Pregnant women not exposed to tildrakizumab

INTERVENTIONS:
Drug: Pregnant women exposed to tildrakizumab — Subjects exposure to tildrakizumab for the treatment of an approved indication, for any number of days, at any dose, and at any time from the first day of the last menstrual period (LMP) up to and including the end of pregnancy
  Groups: Tildrakizumab-Exposed Cohort
Drug: Pregnant women not exposed to tildrakizumab — Subjects diagnosed with a tildrakizumab-approved indication; frequency matched to the exposed group by disease indication, with the indication validated by medical records when possible, and Subjects with no exposure to tildrakizumab at any time in the current pregnancy; may or may not have taken another medication for their disease in the current pregnancy
  Groups: Disease-Matched Comparison Cohort

SUMMARY:
This study will utilize a prospective, observational, exposure cohort design to examine pregnancy and infant outcomes in women and infants who are exposed to tildrakizumab during pregnancy to treat an approved indication.

The pregnancy registry cohort study will be conducted by the Organization of Teratology Information Specialists (OTIS), which is a network of university and health department based information centers serving pregnant women and healthcare providers throughout North America. These services provide a basis for collaborative research such as this Registry.

These Services located throughout the United States (US) and Canada will serve as a source of referrals not only for tildrakizumab-exposed pregnancies but also for similarly ascertained disease-matched comparison pregnant women who have not used tildrakizumab in pregnancy.

The target follow-up period will be until end of pregnancy and 1 year of age for live born infants.

ELIGIBILITY:
Cohort 1: Tildrakizumab-Exposed Cohort

1. Pregnant women
2. Exposure to tildrakizumab for the treatment of an approved indication, for any number of days, at any dose, and at any time from the first day of the last menstrual period up to and including the end of pregnancy
3. Agree to the conditions and requirements of the study including the interview schedule, and release of medical records

Cohort 2: Disease-Matched Comparison Cohort

1. Pregnant women
2. Diagnosed with a tildrakizumab-approved indication; frequency matched to the exposed group by disease indication, with the indication validated by medical records when possible
3. No exposure to tildrakizumab at any time in the current pregnancy; may or may not have taken another medication for their disease in the current pregnancy
4. Agree to the conditions and requirements of the study including the interview schedule, and release of medical records

Exclusion criteria:

Cohort 1: Tildrakizumab-Exposed Cohort:

1. Women who have first contact with the project after prenatal diagnosis of any major structural defect
2. Women who have enrolled in the tildrakizumab cohort study with a previous pregnancy (women may only enroll once in the Tildrakizumab Pregnancy Study)
3. Women who have used tildrakizumab for an indication other than a currently approved indication
4. Retrospective enrollment after the outcome of pregnancy is known

Cohort 2: Disease-Matched Comparison Cohort

1. Women who have first contact with the project after prenatal diagnosis of any major structural defect
2. Exposure to tildrakizumab anytime during the current pregnancy
3. Women who have enrolled in the tildrakizumab cohort study with a previous pregnancy (women may only enroll once in the Tildrakizumab Pregnancy Study)
4. Retrospective enrollment after the outcome of pregnancy is known

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women diagnosed with tildrakizumab-approved indication with and without tildrakizumab
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Major structural defects in children | Up to 1 year of age
  defined and classified using the US Centers for Disease Control and Prevention (CDC) coding manual that is used for the Metropolitan Atlanta Congenital Defects Program (MACDP) classification of major structural defects

SECONDARY OUTCOMES:
Spontaneous abortion/miscarriage | 20 weeks post-last menstrual period
  defined as non-deliberate fetal death that occurs prior to 20.0 weeks post-last menstrual period
Stillbirth | from 20 weeks post-last menstrual period to end of pregnancy
  defined as non-deliberate fetal death anytime in gestation at or after 20.0 weeks post-last menstrual period
Elective termination/abortion | At the end of pregnancy or through 9 month pregnancy period
  defined as deliberate discontinuation of pregnancy through medication or surgical procedures
neonatal/infant death | 6 months of age
  defined as any death in a live born infant during the first 6 months of age
Small for gestational age | at birth
  defined as birth size (weight, length, or head circumference) less than or equal to the 10th centile for sex and gestational age using standard pediatric CDC growth curves for full term or preterm infants
Postnatal growth deficiency | Up to 1 year of age
  defined as postnatal size (weight, length or head circumference) less than or equal to the 10th centile for sex and age using standard pediatric growth curves and adjusted for postnatal age for premature infants if the postnatal measurement is obtained at less than 1 year of age
Malignancies in live born children | Up to 1 year of age
  defined as any malignancy reported in an infant within the first year of life
Hospitalization in live born children | Up to 1 year of age
  defined as any hospitalization of the infant within the first year of life after discharge following delivery
Postnatal serious or opportunistic infection in live born children | Up to 1 year
  defined as any infection resulting in hospitalization, X-ray proven pneumonia, neonatal sepsis, meningitis, osteomyelitis, bacteremia, septic arthritis, abscess, mycobacteria infections, invasive fungal infection including histoplasmosis, coccidiomycosis, candidiasis, aspergillosis, and blastomycosis, pneumocystis jirovecii infection, systemic cytomegalovirus, herpes zoster and herpes simplex infection, listeria infections, and Legionella infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Christina Chambers, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided